CLINICAL TRIAL: NCT01376791
Title: Oral Flora, Periodontitis, and Vascular Dysfunction in Young Native Americans.
Brief Title: Assess the Effect of Treating Periodontal Disease on Cardiovascular Function in Young Adults
Status: Completed | Type: Observational
Sponsor: San Diego State University (Other)
Collaborators: Indian Council of Medical Research (Other Government); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Roberta A. Gottlieb, Director, SDSU BioScience Center, San Diego State University
Other Study IDs: IHC-PDCV
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Periodontal Disease; Atherosclerosis
Keywords: Periodontal disease; Atherosclerosis; Oral Pathogens; Native Americans; Inflammatory cytokines; Microbial metagenomics
MeSH Terms: conditions — Periodontal Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, dental scrapings and saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose to examine a population of Native Americans who have had little or no dental care, and to determine if periodontal disease is associated with early signs of vascular dysfunction or systemic inflammation. We then propose to treat the periodontitis and re-evaluate vascular function. We will determine if gingivitis or mild/moderate periodontitis is associated with detectable vascular dysfunction. Microbial metagenomics will be correlated with vascular function.

ELIGIBILITY:
Inclusion Criteria:

* American Indian/Alaskan Natives seeking health care at the Indian Health Council, Inc.
* Males and females aged 21-40 years.

Exclusion criteria:

* Recent (within 6 months) periodontal treatment
* History of high blood pressure or existing heart disease
* Xerostomia
* Currently receiving treatment for cancer
* Currently taking anti-inflammatory medications (except H2 blockers, statins, or medications that can affect periodontal status
* Immunosuppressed due to medication or HIV infection, or presence of active infection such as hepatitis or tuberculosis
* Fewer than 20 teeth in functional dentition, excluding third molars, or other gross oral pathology

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population comprises 200 Native Americans seeking health care at the Indian Health Council.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determination of bacterial populations in periodontal samples before and after standard periodontal treatment, stratified by severity of gum disease, using microbial metagenomics analysis. | Time of enrollment and at 6 week follow up visit
  The study will assess if periodontal bacterial flora differ in patients with healthy gums, mild, or severe periodontal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A Gottlieb, MD, Principal Investigator — San Diego State University
Locations (1):
- Indian Health Council, Valley Center, California, United States